CLINICAL TRIAL: NCT01928758
Title: Reduced Nicotine Cigarettes in Smokers With Mood and Anxiety Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jonathan Foulds, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY911; P50DA036107 (NIH)
Record Dates: First submitted 2013-08-21; First posted 2013-08-27 (Estimated); Results first posted 2019-02-08 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Tobacco Dependence
Keywords: Smoking; Nicotine
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Nicotine Content Cigarettes (Experimental): The experimental group will smoke cigarettes with gradually Reduced Nicotine Content (11.6, 7.4, 3.3, 1.4, 0.7 and 0.2 mg per cigarette) cigarettes, with each nicotine level smoked for 3 weeks, except the lowest level which continues for 6 weeks
  Interventions: Drug: Reduced Nicotine Content Cigarettes
- Usual Nicotine Content Cigarettes (Placebo Comparator): Research cigarettes with a usual nicotine content (around 11.6mg per cigarette)
  Interventions: Drug: Usual Nicotine Content Cigarettes

INTERVENTIONS:
Drug: Reduced Nicotine Content Cigarettes — Research cigarettes will have gradually reduced nicotine content
  Other Names: Nicotine
  Arms: Reduced Nicotine Content Cigarettes
Drug: Usual Nicotine Content Cigarettes — Usual Nicotine Content Cigarettes
  Other Names: Nicotine
  Arms: Usual Nicotine Content Cigarettes

SUMMARY:
The overall aim of this project is to evaluate the effect of progressive nicotine reduction in cigarettes on smoking behavior, toxin exposure and psychiatric symptoms in smokers with comorbid mood and/or anxiety disorders.

Smokers with mood and/or anxiety disorder will smoke research cigarettes that will contain either a) nicotine content similar to their preferred usual brand of cigarettes, or b) nicotine content per cigarette that is progressively reduced from approximately 11.6 mg to 0.2 mg per cigarette over 18 weeks.

It is our hypothesis that nicotine intake will decline as a function of cigarette nicotine content in the Reduced Nicotine Content group without significant increases in tobacco smoke exposure, severity of nicotine withdrawal symptoms, mood and anxiety symptomatology or protocol non-adherence over time in the Reduced Nicotine Content group as compared with the control group.

DETAILED DESCRIPTION:
The overall aim of this project is to evaluate the effect of progressive nicotine reduction in cigarettes on smoking behavior, toxicant exposure and psychiatric symptoms in smokers with comorbid mood and/or anxiety disorders.

To do so, we will randomly assign 200 adult smokers with a unipolar mood and/or anxiety disorder within the past year to smoke research cigarettes that will contain either a) Usual Nicotine Content (UNC): nicotine content similar to their preferred usual brand of cigarettes, or b) Reduced Nicotine Content (RNC): nicotine content per cigarette is progressively reduced from approximately 11.6 mg to 0.2 mg per cigarette over 18 weeks. All subjects will participate in baseline periods prior to double-blind randomization to assess normal smoking behavior and then to establish ability to tolerate research cigarettes prior to randomization.

A total of 280 participants will be enrolled in the study at two sites with the aim of randomizing 200 who complete the baseline phase. 100 participants will be enrolled in the randomized phase at Penn State Hershey and 100 at the Massachusetts General Hospital site. Participants will be started on the study protocol during Baseline I and Baseline II but will be removed from the study if they are not able to comply with the protocol. We expect that approximately 40 participants at each site drop out from the study prior to randomization (due to inability to comply with study protocol).

It is our hypothesis that nicotine intake, as measured by plasma cotinine concentration, will decline as a function of cigarette nicotine content in the RNC group. Further, it is our hypothesis that by gradually reducing the nicotine content of the cigarettes in a step-wise fashion, there will not be significant increases in biomarkers of tobacco smoke exposure, severity of nicotine withdrawal symptoms, mood and anxiety symptomatology or protocol non-adherence over time in the experimental group (RNC) as compared with the UNC control group.

ELIGIBILITY:
Inclusion Criteria:

* Smoke >4 cigarettes/day for at least a year
* No quit attempt in prior month
* Not planning to quit smoking within next 6 months
* Plan to live in local area for next 8 months
* Meet diagnostic criteria for a current or lifetime Anxiety Disorder or Mood Disorder as determined by the Mini-international Neuropsychiatric Interview
* Read and write in English
* Women not pregnant or nursing and taking steps to avoid pregnancy
* Able to understand and consent to study procedures

Exclusion Criteria:

* Unstable or significant medical condition such as Chronic Obstructive Pulmonary Disease or kidney failure
* Use of non-cigarette nicotine delivery product in the past week or smoking cessation medicine in prior month
* Currently reducing or planning to reduce cigarette consumption in next month
* Uncontrolled serious psychotic illness or substance abuse or inpatient treatment for these in the past 6 months
* Current suicide risk on clinical assessment
* Aged <18 or >65
* History of difficulty providing blood samples (fainting, poor venous access)
* Unwilling to remain on one flavor of cigarette (regular or menthol) for the duration of the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 245 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01-11 (Actual); Study Completion 2018-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan A Foulds, PhD, Principal Investigator — Penn State College of Medicine; A. Eden Evins, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Penn State College of Medicine, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen SI, Foulds J, Pachas GN, Veldheer S, Cather C, Azzouz N, Hrabovsky S, Hameed A, Yingst J, Hammett E, Modesto J, Krebs NM, Zhu J, Liao J, Muscat JE, Richie J, Evins AE. A two-site, two-arm, 34-week, double-blind, parallel-group, randomized controlled trial of reduced nicotine cigarettes in smokers with mood and/or anxiety disorders: trial design and protocol. BMC Public Health. 2017 Jan 19;17(1):100. doi: 10.1186/s12889-016-3946-4. PMID 28103841
- [Derived] Foulds J, Veldheer S, Pachas G, Hrabovsky S, Hameed A, Allen SI, Cather C, Azzouz N, Yingst J, Hammett E, Modesto J, Krebs NM, Lester C, Trushin N, Reinhart L, Wasserman E, Zhu J, Liao J, Muscat JE, Richie JP Jr, Evins AE. The effects of reduced nicotine content cigarettes on biomarkers of nicotine and toxicant exposure, smoking behavior and psychiatric symptoms in smokers with mood or anxiety disorders: A double-blind randomized trial. PLoS One. 2022 Nov 2;17(11):e0275522. doi: 10.1371/journal.pone.0275522. eCollection 2022. PMID 36322562

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 27 participants attended Visit 1 and consented but did not meet final eligibility criteria. The remaining participants (n=218) began a baseline phase during which 30 participants were lost to follow up or withdrawn from the study before being randomized to the study intervention. 188 participants were randomized into an intervention.
Groups:
- Usual Nicotine Content Cigarettes: Research cigarettes with a nicotine content similar to participant's usual brand of cigarettes (around 11.6mg)
  Usual Nicotine Content Cigarettes: Usual Nicotine Content Cigarettes
Period: Overall Study
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Started | 94 | 94
Completed | 69 | 74
Not Completed | 25 | 20
Not completed — Lost to Follow-up | 14 | 9
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Adverse Event | 3 | 5
Not completed — Protocol Violation | 3 | 4

BASELINE CHARACTERISTICS:
Population: Baseline values for outcomes reflect levels after participants were on the usual nicotine content cigarettes for 2 weeks and before they received the intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (11.7) | 43.1 (13.3) | 43.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 54 | 114
  Male | 34 | 40 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 1 | 8
  Not Hispanic or Latino | 87 | 93 | 180
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/white | 70 | 76 | 146
  African American/black | 15 | 11 | 26
  Asian | 1 | 1 | 2
  Native Hawaiian or Pacific Island | 0 | 0 | 0
  American Indian/Alaskan native | 2 | 1 | 3
  Other | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  United States | 94 | 94 | 188
Menthol smoker [Count of Participants; unit: Participants] | 38 | 36 | 74
Quick Inventory of Depressive Symptomatology [Mean (Standard Deviation); unit: units on a scale] — The 16-item scale uses a continuous score and the scale range is 0-27 where 0 = Least Severe and 27 = Most Severe.
  units on a scale | 5.5 (4.8) | 6.3 (4.3) | 5.9 (4.5)
Perceived Stress Scale [Mean (Standard Deviation); unit: units on a scale] — 10-item version was used. Scale range is 0-40. Higher scores indicate more stress.
  units on a scale | 16.0 (7.5) | 17.1 (8.2) | 16.5 (7.9)
Overall Anxiety Severity and Impairment Scale [Mean (Standard Deviation); unit: units on a scale] — The OASIS is a 5-item scale to measure overall anxiety severity and impairment. The range is 0-20 where higher scores indicate higher anxiety.
  units on a scale | 4.9 (4.1) | 5.7 (4.3) | 5.3 (4.2)
Kessler-6 Scale [Mean (Standard Deviation); unit: units on a scale] — The Kessler-6 Scale is a 6-item scale with a total possible score range from 0-24 used to define serious psychological distress. Higher scores indicate more distress.
  units on a scale | 5.6 (5.4) | 6.5 (5.1) | 6.1 (5.3)
Cigarettes per day [Mean (Standard Deviation); unit: cigarettes] | 20.2 (10.7) | 21.6 (10.6) | 20.9 (10.7)
Exhaled Carbon Monoxide [Mean (Standard Deviation); unit: parts per million] | 29.4 (17.7) | 29.1 (15.1) | 29.3 (16.4)
Plasma Cotinine [Mean (Standard Deviation); unit: ng/mL] — Cotinine values below the assay Limit of Detection (LOD) are imputed using a common substitution formula (LOD/ square root of 2), which in the case of plasma cotinine equals 3 ng/mL.
  ng/mL | 245.7 (137.2) | 255.9 (145.5) | 250.9 (141.2)
Minnesota Nicotine Withdrawal Scale [Mean (Standard Deviation); unit: units on a scale] — The scale range is from 0-32 and includes 8 items. The scale is used to measure signs of nicotine withdrawal where higher scores indicate higher severity.
  units on a scale | 9.9 (7.3) | 10.5 (6.3) | 10.2 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Cotinine Concentration
Description: Plasma cotinine is a measure of daily nicotine exposure. Samples were measured in ng/mL.
Time Frame: Measured at the end of the last 3 weeks of randomization trial phase
Population: Randomized trial phase completers with non-missing values for the outcome at both time points being used in the regression (complete case analysis).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 66 | 72
ng/mL | 82.8 (154.3) | 259.0 (151.3)
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Usual Nicotine Content Cigarettes; Test type: Other; p < 0.0001, Regression, Linear — Complete case analysis; Model was adjusted for baseline cotinine after smoking usual nicotine content cigarettes for 2-weeks; Mean Difference (Final Values) = -175.7, 95% CI 2-sided [-218.3 to -133.1] — The direction of comparison is reduced nicotine content vs. usual nicotine content cigarette treatment group

2. Secondary Outcome: Quick Inventory of Depressive Symptomatology
Description: A 16-item scale on depression symptoms. The scale range is 0-27 where 0 = Least Severe and 27 = Most Severe.
Time Frame: Measured at the end of the last 3 weeks of randomization trial phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 69 | 72
score on a scale | 5.5 (4.3) | 5.3 (3.9)
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Usual Nicotine Content Cigarettes; Test type: Other; p = 0.16, Regression, Linear — Complete case analysis; Model was adjusted for baseline score after smoking usual nicotine content cigarettes for 2 weeks; Mean Difference (Final Values) = 0.69, 95% CI 2-sided [-0.28 to 1.65] — The direction of comparison is reduced nicotine content vs. usual nicotine content cigarette treatment group

3. Secondary Outcome: Perceived Stress Scale
Description: 10-item questionnaire measuring the degree to which life situations are appraised stressful. Scale range is 0-40. Higher scores indicate more stress.
Time Frame: Measured at the end of the last 3 weeks of randomization trial phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 69 | 74
score on a scale | 15.0 (7.6) | 15.1 (7.8)
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Usual Nicotine Content Cigarettes; Test type: Other; p = 0.67, Regression, Linear — Complete case analysis; Model was adjusted for baseline score after smoking usual nicotine content cigarettes for 2 weeks; Mean Difference (Final Values) = 0.38, 95% CI 2-sided [-1.40 to 2.16] — The direction of comparison is reduced nicotine content vs. usual nicotine content cigarette treatment group

4. Secondary Outcome: Minnesota Nicotine Withdrawal Scale
Description: This 8-item scale measures nicotine withdrawal symptoms and the scale range is from 0-32. Higher scores indicate higher severity.
Time Frame: Measured at the end of the last 3 weeks of randomization trial phase
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 69 | 74
score on a scale | 8.1 (6.8) | 9.0 (5.9)
Statistical Analysis 1: Comparison: Reduced Nicotine Content Cigarettes vs Usual Nicotine Content Cigarettes; Test type: Other; p = 0.65, Regression, Linear — Complete case analysis; Model was adjusted for baseline score after smoking usual nicotine content cigarettes for 2 weeks; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-1.68 to 1.05] — The direction of comparison is reduced nicotine content vs. usual nicotine content cigarette treatment group

5. Other Pre Specified Outcome: Intention to Quit Smoking
Description: Smokers assigned to the reduced nicotine content cigarette group may have lower perceived dependence and be more likely to report intention to quit smoking
Time Frame: At end of 18-week randomized trial phase
Population: Participants who attended the visit at the end of the 18-week randomized trial phase
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 69 | 74
Participants | 33 | 25

6. Other Pre Specified Outcome: Abstinence From Smoking
Description: Smokers assigned to reduced nicotine content cigarettes will be more likely to successfully abstain from smoking at the end of the trial, based on all randomized participants, defined as no cigarette use in past 7 days, verified by exhaled carbon monoxide <10ppm.
Time Frame: Follow-up appointment 30 weeks after randomization (12 weeks after last visit of randomized trial phase).
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
Number analyzed (Participants) | 94 | 94
Participants | 17 | 4

ADVERSE EVENTS:
Time Frame: All randomized participants throughout the entire 33 weeks of the trial.
Description: Adverse events (AEs) were systematically collected at each study visit by asking participants about any changes in their physical or mental health or if they needed to seek immediate medical care at an emergency room or hospital.
Groups:
- Reduced Nicotine Content Cigarettes: The experimental group will smoke cigarettes with gradually Reduced Nicotine Content (11.6, 8.6, 4.0, 1.8, 0.9 and 0.3 mg per cigarette) cigarettes, with each nicotine level smoked for 3 weeks, except the lowest level which continues for 6 weeks
  Reduced Nicotine Content Cigarettes: Research cigarettes will have gradually reduced nicotine content
Arm/Group | Reduced Nicotine Content Cigarettes | Usual Nicotine Content Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/94
Serious Adverse Events (participants affected / at risk) | 7/94 | 10/94
Other Adverse Events (participants affected / at risk) | 70/94 | 72/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Nicotine Content Cigarettes (N=94) | Usual Nicotine Content Cigarettes (N=94)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0) — Blocked artery
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Endocarditis infective (Infections and infestations) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 1 (1) — Lung and leg infection
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Accidental drug overdose
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Rhabdomyolysis
Psychiatric disorders - Other (Psychiatric disorders) | 0 (0) | 1 (1) — Drug relapse
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 0 (0) | 1 (1) — Dog bite requiring surgery
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reduced Nicotine Content Cigarettes (N=94) | Usual Nicotine Content Cigarettes (N=94)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Anxiety (Psychiatric disorders) | 22 (28) | 19 (22)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5)
Depression (Psychiatric disorders) | 30 (39) | 21 (26)
Flu like symptoms (General disorders) | 9 (9) | 11 (14)
Headache (Nervous system disorders) | 8 (9) | 4 (5)
Hypertension (Vascular disorders) | 3 (3) | 7 (7)
Irritability (Psychiatric disorders) | 4 (4) | 6 (7)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 9 (13) | 13 (15)
Suicidal ideation (Psychiatric disorders) | 14 (14) | 11 (11)
Surgical and medical procedures - Other (Surgical and medical procedures) | 5 (5) | 5 (5)
Upper respiratory infection (Infections and infestations) | 29 (32) | 24 (30)

LIMITATIONS AND CAVEATS:
The sample size was not reached due to a shortage of study cigarette inventory.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT01928758/Prot_SAP_000.pdf